CLINICAL TRIAL: NCT02023333
Title: Phase II Study of Regorafenib in Good Performance Status Patients With Newly Diagnosed Metastatic Colorectal Adenocarcinoma
Brief Title: Regorafenib in Good Performance Status Patients With Newly Diagnosed Metastatic Colorectal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry); State University of New York - Downstate Medical Center (Other); Queens Cancer Center of Queens Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-211
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Colorectal Adenocarcinoma
Keywords: Regorafenib; Performance Status; 13-211
MeSH Terms: interventions — regorafenib

ARMS (1):
- Regorafenib (Experimental): This is an open-label, phase II study of regorafenib for patients with metastatic colorectal carcinoma. The treatment will be repeated every week for three weeks on and one week off. Patients will be evaluated for response after every 2 cycles (8 weeks).
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — All patients that meet the eligibility criteria who have signed informed consent and have enrolled on the trial will be treated with regorafenib, daily 3 weeks on 1 week off for all cycles. Dose will be escalated to 120 mg in week 2 of cycle 1 and all remaining cycles if no excess toxicity is experienced by the patient at the discretion of the treating physician.
  Other Names: BAY 73-45060

SUMMARY:
The purpose of this study is to evaluate the good and bad effects when regorafenib is used instead of standard combination chemotherapy. It is not known if taking regorafenib versus standard chemotherapy will have better, worse or the same results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Life expectancy of at least 12 weeks (3 months).
* Untreated for metastatic colorectal cancer, or progression on any first line 5-FU containing regimen (such as FOLFOX or FOLFIRI)
* Histologically proven colorectal adenocarcinoma

  * Metastatic disease, unresectable disease involving one or more sites including liver, lung, lymph nodes and peritoneum, with each nodule measuring ≤3cm OR no more than two sites of disease (two nodules) >4.5 cm.
* ECOG 0 or 1
* Adequate bone marrow, liver and liver function as assessed by the following laboratory requirements:
* Total bilirubin ≤ 1.5 x the upper limits of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 xULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
* Alkaline phosphastase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
* Lipase ≤ 1.5 x the ULN
* Creatinine ≤ 1.5 x the ULN
* Platelet count ≥ 100000 /mm3
* hemoglobin (Hb) ≥ 9 g/dL,
* absolute neutrophil count (ANC) ≥ 1500/mm3.
* Blood transfusion to meet the inclusion criteria will not be allowed.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 3 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the site principal investigator or a designated associate.
* Subject must be able to swallow and retain oral medication.
* If the patient is enrolled at MSK he/she must consent to a pre and post treatment biopsy (or have archived tissue available for the pretreatment analysis). Pretreatment archival tissue for patients enrolled outside of MSK should be submitted to MSK. If there is no archival tissue available, a repeat biopsy is not required for non-MSK patients.

Exclusion Criteria:

* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease including:
* Congestive heart failure - New York Heart Association (NYHA) > Class II.
* Active coronary artery disease.
* Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
* Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or
* Recent history of prior cancer except cervical cancer in situ, treated basal cell carcinoma, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before enrollment are allowed.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Ongoing infection > Grade 2 NCI-CTCAE v4.0.
* Symptomatic metastatic brain or meningeal tumors.
* Presence of a non-healing wound, non-healing ulcer, or bone fracture.
* Patients with seizure disorder requiring medication.
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 4.0 Grade 2 dyspnea).
* History of organ allograft (including corneal transplant).
* Any malabsorption condition.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
progression free survival | 16 weeks
  Response and progression will be evaluated in this study using the international criteria proposed by the RECIST 1.1 Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria.

SECONDARY OUTCOMES:
overall survival | 2 years
  Overall survival is defined as the time from treatment start to death or last follow up. Survival will be estimated using the Kaplan-Meier method.
disease control rate | 16 weeks
  Disease control rate (defined with RECIST 1.1 criteria at 16 weeks (2nd scan) as CR, PR or SD), will be estimated using proportions and exact binomial 95% confidence intervals provided.
duration of stable disease | 2 years
  Duration of stable disease will be defined as the time from stable disease to the time of documented progression.
toxicity | 2 years
  will be evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.0. The assessments will be based on recorded adverse events, physical examinations, and clinical laboratory assessments. Toxicity will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Downstate Medical Center, Brooklyn, New York
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center Sleepy Hollow, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/